CLINICAL TRIAL: NCT03880396
Title: Definitive Concurrent Hypofractionated Radiotherapy With Weekly Cisplatin in Locally Advanced Squamous Cell Carcinoma Head and Neck (SCCHN)
Brief Title: Definitive Concurrent Hypofractionated Rth With Weekly Cisplatin in Locally Advanced SCCHN
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Doaa Gamal Abdelnaser Fathy Mahmoud, Principle investigator, Assiut University
Other Study IDs: chemoradiation in SCCHN
Record Dates: First submitted 2018-07-06; First posted 2019-03-19 (Actual); Last update posted 2022-07-26 (Actual); Status verified 2022-07

CONDITIONS: Squamous Cell Carcinoma of the Head and Neck
Keywords: chemoradiation, IMRT, Head and neck cancer
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Head and Neck Neoplasms | interventions — Cisplatin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- hypofractionated Rth with weekly cisplatin 40mg/m2: hypofractionated radioyherapy with weekly cisplatin 40mg/m2
  Interventions: Radiation: hypofractionated Rth with platinol

INTERVENTIONS:
Radiation: hypofractionated Rth with platinol — hypofractionated Rth with weekly cisplatin 40mg/m2

SUMMARY:
The primary endpoint will be acute toxicity. Secondary endpoints included: late toxicity and quality of life; loco-regional control, disease free survival and overall survival.

DETAILED DESCRIPTION:
Head and neck cancer is considered the 6th most common cancer all over the world, with 890,000 new cases and 450,000 deaths in 2018 (1). The histologic type in more than 90% of head and neck cancer is squamous cell carcinoma (SCC) (2). The incidence of SCC in head and neck (SCCHN) continues to rise and is expected to increase by 30% in 2030, which means about 1.08 million new cases annually (3). Hospital-based studies in Egypt showed that SCCHN represents about 20% of all malignancies. The overall incidence of SCCHN in Egypt from 1999 to 2006 was approximately twice among males (476,000) than in females (273,000) (4). Males are affected significantly more than females, with a ratio ranging from 2:1 to 4:1 (5).

Tobacco and alcohol consumption are the high-risk factors of SCCHN (6). Human papilloma virus (HPV), especially subtypes 16 and 18 are implicated risk factors in oropharyngeal cancer (7). Some studies found an association between HPV and P53 gene mutation, as HPV expresses two viral proteins (E6 and E7 proteins) that inactivates P53 and pRB genes, causing genomic instability and malignant transformation ((8)). SCCHN arises from the mucosal epithelium of the oral cavity, nasopharynx, oropharynx, hypopharynx, and larynx. HPV associated SCCHN arises primarily from the palatine and lingual tonsils of the oropharynx, whereas tobacco associated SCCHN arises primarily in the oral cavity, hypopharynx, and larynx.

SCCHN is being increasingly treated by multimodality approaches combining surgery, radiotherapy (RT), and chemotherapy (CTH). Randomized controlled trials have demonstrated major improvements in loco-regional tumor control (LRC) from altered fractionation RT with CTH as compared with conventional fractionated RT (CFRT) (9). Altered fractionation schedules reduces tumor repopulation effect and seek to improve the therapeutic ratio between tumor cell killing and normal tissue damage. Additionally, some data showed that cancer patients are at higher risk of COVID-19 infection comparing with the general population due to many treatment visits, so hypo-RT schedules are better for these patients. hypo-RT utilizes a small number of fractions with a larger dose per fraction (> 2Gy per fraction), shortening overall treatment time compared to a CFRT (9). Although a shorter treatment time can be obtained by applying a higher dose per fraction, it might also result in an increase in the incidence of late complications.

The aim of this study was to investigate hypo fractionated intensity modulated RT (hypo-IMRT) with 62.5 Gy in 25 daily fractions over five weeks (2.5 Gy per fraction with weekly cisplatin 40mg/m2 in patients with high-risk stage II (T2N0, excluding glottic laryngeal) disease, stage III (T1-3 N1 or T3N0) and stage IV (T1-4N2 orN3). The primary endpoint will be assessment of acute toxicity. Secondary endpoints included: late toxicity and quality of life; LRC, disease free survival (DFS) and overall survival (OS).

ELIGIBILITY:
Inclusion Criteria:

* Have histologically or cytologically proven oropharyngeal, laryngeal or hypopharyngeal squamous cell carcinoma; with AJCC high risk stage II (T2N0, excluding glottic laryngeal) disease, stage III (T1-3N1 or T3N0) and stage IV (T1-4N2 or N3) Locally advanced non metastatic stage II/IV SCCHN according to AJCC stage classification 2018 (8th edition);
* Age >18 years and <75 years;
* No previous treatment(neither chemotherapy nor radiotherapy);
* Eastern Cooperative Oncology Group(ECOG) performance status of <2;
* Adequate organ function;
* Provide informed oral or written consent.

Exclusion Criteria:

* prior surgical curative resection for primary tumor;
* patients with metastatic disease;
* prior radiotherapy within the treatment field;
* any relative contraindication to radiotherapy;
* prior administration of EGFR monoclonal antibodies, signal transduction inhibitors or targeted therapies;
* Active severe infection;
* Active concomitant malignancy;
* Pregnant and or lactating women;
* Pre-existing motor or sensory neurotoxicity > CTCAE grade 2.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A planned 62 patients were recruited in the period from 2018 to 2021, 52(83.9%) were males and the remaining 10 (16.1%) were females. 22 of patients were current smoker. Patients had histologically or cytologically proven oropharyngeal (32.3%), laryngeal (32.3%) or hypopharyngeal squamous cell carcinoma (18.2%); with AJCC high risk stage II (T2N0, excluding glottic laryngeal) disease (22.6%), stage III (T1-3N1 or T3N0) (30.6%) and stage IV (T1-4N2 or N3) (46.8%). Human papilloma virus status was not tested at the time of paper design.
Sampling Method: Non-Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2019-03-10 (Actual); Primary Completion 2020-12-26 (Actual); Study Completion 2020-12-26 (Actual)

PRIMARY OUTCOMES:
number of patients havingdegrees of Number of patients having acute toxicities of hypofractionated radiotherapy ,Number of patients with locoregional recurrence-free interval | 2 years
  degree of acute toxicity (mucosititis degree) according to RECIST criteria,degree of dysphagia ,Number of patients with locoregional recurrence-free interval This is assessed by imaging studies and/or physical exams at follow- up visits. This will include a diagnostic FDG PET/CT scan. CT and/or MRI of the primary site and neck will also be recommended. Patients will be classified as locoregional recurrence-free as long as there is no evidence of locoregional recurrence of disease by clinical evaluation, CT, MRI, and/or PET-CT according to the standard of care. For patients achieving complete response of disease, no further imaging study is necessary.

SECONDARY OUTCOMES:
number of patients having degrees of late toxicities of chemoradiation, disease free survival interval,overall survival interval | 2 years
  number of patients having late toxicity (grade's of xerostomia, dysphagia), disease free survival, overall survival accordind to RECIST criteria This is assessed by imaging studies and/or physical exams at follow- up visits. This will include a diagnostic FDG PET/CT scan. CT and/or MRI of the primary site and neck will also be recommended. Patients will be classified as disease-free survival as long as there is no evidence of locoregional recurrence of disease by clinical evaluation, CT, MRI, and/or PET-CT according to the standard of care. For patients achieving complete response of disease, no further imaging study is necessary.
Disease free survival, overall survival, locoregional control | 2 year
  to detect the 2y-DFS,2y-OS,

CONTACTS AND LOCATIONS:
Overall Officials: Doaa G Abdelnaser Fathy Mahmoud, Doctor, Principal Investigator — Assiut University; Hoda H Essa, Doctor, Principal Investigator — Assiut University; Aiat M Mohammed, Doctor, Principal Investigator — Assiut University; Mohamed O Gad, Doctor, Principal Investigator — Assiut University; Nora Essam, Principal Investigator — South Egypt Cancer Institute
Locations (1):
- Assiut university, Asyut, Egypt

REFERENCES:
- [Result] Thomson DJ, Ho KF, Ashcroft L, Denton K, Betts G, Mais KL, Garcez K, Yap BK, Lee LW, Sykes AJ, Rowbottom CG, Slevin NJ. Dose intensified hypofractionated intensity-modulated radiotherapy with synchronous cetuximab for intermediate stage head and neck squamous cell carcinoma. Acta Oncol. 2015 Jan;54(1):88-98. doi: 10.3109/0284186X.2014.958528. Epub 2014 Oct 3. PMID 25279959
- [Result] Szutkowski Z, Kawecki A, Jarzabski A, Laskus Z, Krajewski R, Michalski W, Kukolowicz P. Hypofractionated accelerated radiotherapy in T1-3 N0 cancer of the larynx: A prospective cohort study with historical controls. Rep Pract Oncol Radiother. 2016 Nov-Dec;21(6):537-543. doi: 10.1016/j.rpor.2016.08.001. Epub 2016 Sep 20. PMID 27698593
- See also: Hypofractionated accelerated radiotherapy in T1-3 N0 cancer of the larynx: A prospective cohort study with historical controls. Rep Pract Oncol Radiother. 2016 Nov-Dec — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC5035337/

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-07-20): https://cdn.clinicaltrials.gov/large-docs/96/NCT03880396/Prot_SAP_000.pdf